CLINICAL TRIAL: NCT04159792
Title: Factors Influencing on Postural Balance and Voluntary Movement in Individuals With Acute Stroke
Brief Title: Factors Influencing Postural Balance and Movement in Individuals With Stroke
Acronym: FIPBMS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Vimonwan Hiengkaew (Other)
Responsible Party: Sponsor-Investigator, Vimonwan Hiengkaew, Principle investigator, Mahidol University
Organization: Mahidol University (Other)
Other Study IDs: 2019/199.3007
Record Dates: First submitted 2019-11-06; First posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Stroke; Movement, Abnormal; Postural, Balance
Keywords: stroke; upper limb; lower limb; mobility; posture
MeSH Terms: conditions — Stroke; Dyskinesias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- stroke: Those with standard treatment as usual.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — No intervention

SUMMARY:
There are several factors influencing on balance and movement in individuals with stroke, such as previous stroke, age, bowel incontinence, visuospatial problem. However, those factors involving in postural control and voluntary movement were studied in subacute and chronic phase of stroke, but not in the acute period. The aim of the study is to determine factors for postural control and voluntary movement in individuals with acute stroke and then follow at the first, third, and sixth month.

DETAILED DESCRIPTION:
Background

Postural control is an important component of movement. Prior to movement initiation, it is necessary to control posture such as gait initiation. Individuals with stroke often show impairment in both postural control and voluntary movement. The deficiencies restrict individuals with stroke to perform activities daily living and reduce quality of life leading to a great burden on family members and healthcare system. Additionally, there are positive association between postural control and movement. Therefore, postural control influences movement in individuals with stroke that may be in long term.

Factors influencing on postural control and voluntary movement are shown in subacute and chronic phase of stroke. Previous stroke, age, bowel incontinence, visuospatial problem, initial severe hemiplegia, lesion edema, and intraparenchymal bleeding can predict postural control. Static and dynamic postural balance can predict functional outcome and discharge destination, as well as independent ambulation in individuals with stroke. Level of paresis, motor-evoked potentials, and size of lesion can predict voluntary movement. Furthermore, baseline upper extremity (UE) voluntary movement, hemorrhagic stroke, baseline National Institutes of Health Stroke Scale (NIHSS), and cortical lesion excluding primary motor cortex can predict outcome of UE movement in subacute stroke. Admission lower extremity (LE) voluntary movement score and volume and edema of lesion are predictors for motor recovery of LE at discharge from rehabilitation ward. Age, severity of LE weakness, visual problems, size of lesion, and type of stroke are predictors for walking ability within 30 days after stroke.

Those factors associating with postural control and voluntary movement were studied in subacute and chronic phase of stroke, but not in the acute period. The findings may limit to apply to the earlier period of stroke since different mechanisms of recovery occurring in different timing after brain injury. Additionally, in clinical practice, one of the common questions that clinicians are often asked by individuals with stroke and family members is whether he/she can sit, stand, and walk. To provide an assurance response, the factors associated with postural control and voluntary movement in the acute phase of stroke is required.

Furthermore, previous studies investigating predictors of postural control and voluntary movement used diverse outcome measures. Posture control were examined by different measures, for example Barthel Index, Mini-Mental State Examination, Frenchay Activity Index and Rankin Scale. Similarly, motor function recovery was assessed by various outcomes such as Scandinavian Stroke Scale, Medical Research Council scale, Motricity index, and exclusive of own scale. These measurements indirectly assessed postural control and voluntary movement. However, there is a measure directly examining postural control and voluntary movement for individuals with stroke that is Postural Assessment Scale for Stroke (PASS) and Stroke Rehabilitation Assessment of Movement (STREAM). These two measurements have excellent reliability and show no floor or ceiling effect in acute stroke. In addition, the PASS is an outcome measure recommended for acute stroke care. It would be, therefore, better using PASS and STREAM to record and for communication.

The aim of the study is to determine factors for postural control and voluntary movement in individuals with acute stroke and then follow at the first, third, and sixth month.

Methods

The study is observation clinical research. Participants are individuals with stroke admitted to acute stroke unit, Siriraj hospital. They are included if they are first stroke and aged 18 years and over. They are excluded if they recurrent stroke, have other neurological diseases such as brain tumor, Parkinson's Disease, systolic blood pressure greater than 160 mmHg and/or diastolic blood pressure greater than 100 mmHg, heart failure recorded in patient's file, joint limitation in functional range, and difficulty in communication (i.e. sensory aphasia, severe hearing loss). The sample size is calculated with 15% dropout and requires 103 participants.

A researcher will contact physical therapist who is on duty to ask for patients who are in the inclusion criteria. Then, a researcher contacts patients or family members taking responsibility for patients via face to face to inform the study and ask he/she to sign written inform consent if he/she would like to participate in the study. Within 3 days of admission, a researcher will extract the information from patients' file. The information is age, gender, body mass index, Glasgow coma score, onset to admission interval (OAI), hemisphere lesion, affected side, initial National Institute Health Stroke Scale (NIHSS-IN), history of receiving recombinant tissue plasminogen activator (rtPA), thrombectomy, craniotomy, craniectomy, receiving transcranial direct current stimulation (tDCS), days staying in acute stroke unit (DOS), days from admission to first physical therapy (DA-PT), days receiving physical therapy (DPT), days from baseline to final assessment (D-B-FA). Furthermore, progressive stroke and physical therapy treatments are noted. Additionally, the researcher will assess postural control by PASS and voluntary movement by STREAM that will be baseline PASS (PASS-B) and baseline STREAM (STREAM-B). The researcher will take NIHSS score of that day from patient's file (NIHSS-B). The PASS-B includes baseline score of ability to maintain posture (PASS-B_M) and baseline score of ability to control balance changing position (PASS-B_C). The STREAM-B consists of score of upper extremity movement (STREAM-B_UE), baseline score of lower extremity movement (STREAM-B_LE), and baseline score of basic mobility (STREAM-B_Mo).

Before 2 days of discharge or on the day of discharge from the ward the same researcher will assess postural control and voluntary movement again. Hence, the data will be PASS at discharge (PASS-DC) and its subitems (PASS-DC_M; PASS-DC_C), STREAM at discharge (STREAM-DC) and its subitems (STREAM-DC_UE; STREAM-DC_LE; STREAM-DC_Mo).

After discharge at 1st, 3rd, and 6th month participants will assess postural control (PASS-1, PASS-3, PASS-6) and its subitems (PASS-1_M, PASS-1_C, PASS-3_M; PASS-3_C, PASS-6_M; PASS-6_C) voluntary movement (STREAM-1, STREAM-3, STREAM-6) and its subitems (STREAM-1_UE; STREAM-1_LE; STREAM-1_Mo, STREAM-3_UE; STREAM-3_LE; STREAM-3_Mo, STREAM-6_UE; STREAM-6_LE; STREAM-6_Mo). Participants will be contacted via phone to make an appointment for the assessment at Siriraj hospital or home depending on convenience of participants.

Descriptive analysis is performed for subject characteristics with frequency or mean and SD, as appropriate. Association between any of continuous or categorical variables and NIHSS-DC, PASS-DC, STREAM-DC, PASS-1, STREAM-1, PASS-3, STREAM-3, PASS-6, or STREAM-6 is conducted by Pearson correlation or Spearman correlation test, as appropriate. To identify the potential factors for postural control and voluntary movement, univariate analysis is conducted for all variables, then followed by the regression analysis. If the association shows significance with p-value < 0.05, the candidate variable can be assumed as potential factor. Finally, a multiple linear regression analysis was performed to determine the last predictors for PASS and STREAM at discharge. Multicollinearity among independent factors is tested by variance inflation factor (VIF) and admitted if VIF > 10.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old and over
2. First stroke

Exclusion Criteria:

1. Recurrent stroke
2. Having other neurological diseases such as brain tumor, Parkinson's Disease
3. Systolic blood pressure greater than 160 mmHg and/or diastolic blood pressure greater than 100 mmHg
4. Having heart failure recorded in patient's file
5. Having joint limitation in functional range
6. Difficulty in communication (i.e. sensory aphasia, severe hearing loss)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with stroke.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Estimated)
Dates: Start 2019-11-10 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2022-11-09 (Estimated)

PRIMARY OUTCOMES:
National Institutes of Health Stroke Scale | 6 months
  severity of stroke
Postural Assessment Scale for Stroke | 6 months
  postural balance
Stroke Rehabilitation Assessment of Movement | 6 months
  voluntary movement

SECONDARY OUTCOMES:
subitem of Postural Assessment Scale for Stroke | 6 months
  maintain and change posture
subitem of Stroke Rehabilitation Assessment of Movement | 6 months
  upper and lower limb movement and basic mobility

CONTACTS AND LOCATIONS:
Overall Officials: Vimonwan Hiengkaew, PhD, Principal Investigator — Faculty of Physical Therapy, Mahidol University
Locations (1):
- Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ivanenko Y, Gurfinkel VS. Human Postural Control. Front Neurosci. 2018 Mar 20;12:171. doi: 10.3389/fnins.2018.00171. eCollection 2018. PMID 29615859
- [Background] Hass CJ, Gregor RJ, Waddell DE, Oliver A, Smith DW, Fleming RP, Wolf SL. The influence of Tai Chi training on the center of pressure trajectory during gait initiation in older adults. Arch Phys Med Rehabil. 2004 Oct;85(10):1593-8. doi: 10.1016/j.apmr.2004.01.020. PMID 15468016
- [Background] Skolarus LE, Burke JF, Brown DL, Freedman VA. Understanding stroke survivorship: expanding the concept of poststroke disability. Stroke. 2014 Jan;45(1):224-30. doi: 10.1161/STROKEAHA.113.002874. Epub 2013 Nov 26. PMID 24281223
- [Background] Rajachandrakumar R, Fraser JE, Schinkel-Ivy A, Inness EL, Biasin L, Brunton K, McIlroy WE, Mansfield A. Atypical anticipatory postural adjustments during gait initiation among individuals with sub-acute stroke. Gait Posture. 2017 Feb;52(1):325-331. doi: 10.1016/j.gaitpost.2016.12.020. Epub 2016 Dec 21. PMID 28038342
- [Background] Craig LE, Wu O, Bernhardt J, Langhorne P. Predictors of poststroke mobility: systematic review. Int J Stroke. 2011 Aug;6(4):321-7. doi: 10.1111/j.1747-4949.2011.00621.x. PMID 21745343
- [Background] Huang YC, Wang WT, Liou TH, Liao CD, Lin LF, Huang SW. Postural Assessment Scale for Stroke Patients Scores as a predictor of stroke patient ambulation at discharge from the rehabilitation ward. J Rehabil Med. 2016 Mar;48(3):259-64. doi: 10.2340/16501977-2046. PMID 26667386
- [Background] Daley K, Mayo N, Wood-Dauphinee S. Reliability of scores on the Stroke Rehabilitation Assessment of Movement (STREAM) measure. Phys Ther. 1999 Jan;79(1):8-19; quiz 20-3. PMID 9920188
- [Background] Lesser M BJ, Dekerlegand J. Use of the postural assessment scale for stroke patients in determining acute care discharge recommendations. J Acute Care Phys Ther 2017:79-85.